CLINICAL TRIAL: NCT00279487
Title: Preanalgesic Effect of Gabapentin in Total Knee Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Health Resources (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P768
Record Dates: First submitted 2006-01-16; First posted 2006-01-19 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Patients undergoing total knee replacement who received pain management by the following modality:; IV PCA opioid; Local femoral nerve block with 1.5% Mepivacaine & 0.5% Ropivacaine
MeSH Terms: conditions — Pain | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Patients will receive 1200mg gabapentin 1-2 hours prior to surgery.
  Interventions: Drug: Gabapentin
- Arm 2 (Placebo Comparator): Patients will receive placebo 1-2 hours prior to surgery.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Gabapentin
  Arms: Arm 1
Drug: Placebos
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine whether gabapentin, as a one time administration prior to a total knee replacement procedure, has opioid sparing effects and a reduction in pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee replacement who received pain management by the following modality:

  * Intravenous patient-controlled analgesia (IV-PCA) opioid
  * Local femoral nerve block with 1.5% mepivacaine 20 ml and 0.5% ropivacaine 20 ml

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob Hutchison, Principal Investigator — Texas Health Resources
Locations (1):
- Presbyterian Hospital of Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No